CLINICAL TRIAL: NCT01490580
Title: Double Blind Randomized Controlled Trial Comparing "Atropine+Propofol" Versus "Atropine+Atracurium+Sufentanil" as a Premedication Prior to Semi-urgent or Elective Endotracheal Intubation of Term and Preterm Newborns
Brief Title: Premedication Trial for Tracheal Intubation of the NEOnate
Acronym: PRETTINEO
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Collaborators: Association Clinique Thérapeutique Infantile du val de Marne (Other)
Responsible Party: Principal Investigator, Xavier Durrmeyer, Principal Investigator, Centre Hospitalier Intercommunal Creteil
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRETTINEO
Record Dates: First submitted 2011-12-08; First posted 2011-12-13 (Estimated); Results first posted 2019-09-13 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-02

CONDITIONS: Premedication; Endotracheal Intubation
Keywords: Pain; Newborn; Anaesthesia; opioids; propofol; neuromuscular blocker; atropine
MeSH Terms: conditions — Pain | interventions — Atropine; Atracurium; Sufentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atropine + Propofol (Experimental)
  Interventions: Drug: atropine+ propofol
- Atropine + atracurium + sufentanil (Active Comparator)
  Interventions: Drug: atropine + atracurium + sufentanil

INTERVENTIONS:
Drug: atropine+ propofol — Atropine bolus: 20 µg/kg Propofol injected over 60 seconds: 1 mg/kg for infants < 1000g - Renewable once 2.5 mg/kg for infants > 1000G - Possible additional dose of 1 mg/kg
  Arms: Atropine + Propofol
Drug: atropine + atracurium + sufentanil — Atropine bolus: 20 µg/kg Atracurium: 0.3 mg/kg- Possible additional dose of 0.1 mg/kg Sufentanil: 0.1 µg/kg for infants < 1000g 0.2 µg/kg for infants > 1000g
  Arms: Atropine + atracurium + sufentanil

SUMMARY:
Multicenter double blind randomized controlled trial comparing "atropine+propofol" vs "atropine+atracurium+sufentanil" as a premedication prior to endotracheal intubation of the neonate.

Primary outcome: pulse oxymetry value < 80% for more than 60 seconds. Secondary outcomes: number of attempts, duration of the procedure, changes in physiologic parameters, short- and long-term neurodevelopmental outcome.

Hypothesis: "atropine + propofol" compared to "atropine+atracurium+sufentanil" will significantly reduce the frequency of severe hypoxemia.

ELIGIBILITY:
Inclusion Criteria:

* Corrected age < 45 weeks of gestational age
* Currently hospitalized in a neonatal intensive care unit
* Requiring semi-urgent or elective intubation
* Equipped with a reliable and permeable IV line
* Parental consent

Exclusion Criteria:

* Lack of parental consent
* Parental refusal
* Sedative or anesthetic treatment in the previous 24 hours
* Hemodynamic compromise defined as mean blood pressure< corrected GA and/or refill time > 3 seconds
* Upper airway malformation
* Life-threatening situation requiring immediate intubation
* Inclusion in another trial not permitting any other participation
* Impossibility to establish venous access
* Any contra-indication to any experimental drug

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 173 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2020-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Durrmeyer, MD, Principal Investigator — CHI CRETEIL
Locations (6):
- France (6):
  - Médecine Néonatale et Réanimation Pédiatrique Polyvalente, CHU Amiens Nord, Amiens
  - Hôpital Mère-Enfant, Bron
  - CHU de Caen, Caen
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - Hôpital des Enfants, Toulouse
  - Réanimation Pédiatrique et Néonatale de l'hôpital Clochevile, Centre Hospitalier Universitaire de Tours, Tours

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Durrmeyer X, Breinig S, Claris O, Tourneux P, Alexandre C, Saliba E, Beuchee A, Jung C, Levy C, Marchand-Martin L, Marcoux MO, Dechartres A, Danan C; PRETTINEO Research Group. Effect of Atropine With Propofol vs Atropine With Atracurium and Sufentanil on Oxygen Desaturation in Neonates Requiring Nonemergency Intubation: A Randomized Clinical Trial. JAMA. 2018 May 1;319(17):1790-1801. doi: 10.1001/jama.2018.3708. PMID 29715354
- [Result] Tauzin M, Marchand-Martin L, Lebeaux C, Breinig S, Claris O, Tourneux P, Alexandre C, Levy C, Jung C, Dechartres A, Durrmeyer X; PREmedication Trial for Tracheal Intubation of the NEOnate Research Group. Neurodevelopmental Outcomes after Premedication with Atropine/Propofol vs Atropine/Atracurium/Sufentanil for Neonatal Intubation: 2-Year Follow-Up of a Randomized Clinical Trial. J Pediatr. 2021 Apr;231:273-277.e3. doi: 10.1016/j.jpeds.2020.12.001. Epub 2020 Dec 8. PMID 33301785

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was prematurely interrupted for logistic reasons in July 2016: a fourth drug manufacturing run was necessary because the intralipids had passed their expiration date and funding had run out. During the study period, 755 patients were screened for eligibility, and 173 randomized
Groups:
- Atropine Atracurium Sufentanil: n=82 allocated to atropine+atracurium+sufentanil
  * n=80 received allocated intervention
  * n=2 did not receive allocated intervention
  * n=1 never intubated
  * n=1 received another premedication
    82 included in final analysis
- Atropine Propofol: n=91 allocated to atropine+propofol
  * n= 2 excluded for lack of consent
  * n=83 received allocated intervention
  * n=6 did not receive allocated intervention
  * n=2 never intubated
  * n=4 received another premedication
    89 included in final analysis
Period: Overall Study
Arm/Group | Atropine Atracurium Sufentanil | Atropine Propofol
Started | 82 | 91
Completed | 82 | 89
Not Completed | 0 | 2
Not completed — Parents withdrew consent | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atropine Atracurium Sufentanil | Atropine Propofol | Total
Number analyzed (Participants) | 82 | 89 | 171
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 82 | 89 | 171
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: days] | 1 [0 to 10] | 1 [0 to 9] | 1 [0 to 10]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 45 | 70
  Male | 57 | 44 | 101
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 82 | 89 | 171
Median GA at birth [IQR], weeks [Median (Inter-Quartile Range); unit: WEEKS] | 29 [26 to 32] | 30 [28 to 34] | 29 [27 to 33]
Median birth weight [IQR], g [Median (Inter-Quartile Range); unit: GRAMS] | 1130 [850 to 1685] | 1310 [815 to 2385] | 1190 [830 to 2020]
Reason for intubation, n (%) [Count of Participants; unit: Participants]
  Respiratory distress syndrome | 50 | 60 | 110
  Apnea | 9 | 3 | 12
  Surgery | 16 | 20 | 36
  Other | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Prolonged Desaturation
Description: Pulse oxymetry value measured by Masimo technology below 80% for 60 seconds or more.
  Duration of intubation is defined by the time between first laryngoscope insertion and last laryngoscope removal after successful intubation. Successful intubation is defined by clear bilateral breath sounds, increasing heart rate and saturation (if previously low) and appropriate flow curves on the ventilator.
Time Frame: During intubation procedure, expected duration 1 to 15 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Atropine Atracurium Sufentanil | Atropine Propofol
Number analyzed (Participants) | 82 | 89
Participants | 54 | 53
Statistical Analysis 1: Comparison: Atropine Atracurium Sufentanil vs Atropine Propofol; Test type: Superiority; p = 0.38, Mixed Models Analysis; Risk Difference (RD) = -6.4, 95% CI 2-sided [-21.0 to 8.1]

2. Secondary Outcome: Number of Intubation Attempts
Time Frame: During intubation procedure, expected duration 1 to 15 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Atropine + Propofol | Atropine + Atracurium + Sufentanil
Number analyzed (Participants) | 89 | 82
Participants
  1 attempt | 41 | 47
  2 attempts | 25 | 23
  > 2 attempts | 21 | 11
  Missing data | 2 | 1

3. Secondary Outcome: Duration of Intubation Procedure
Description: Although the initial definition of procedure duration in the registered protocol was the time between the first laryngoscope insertion and last laryngoscope removal after successful intubation, the variable collected in the clinical research form was defined as the time between first laryngoscope insertion and the fixation of the tube with tape.
Time Frame: Expected duration 1 to 15 minutes
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Atropine + Propofol | Atropine + Atracurium + Sufentanil
Number analyzed (Participants) | 84 | 80
Minutes | 6.0 [2.8 to 9.1] | 3.5 [1.3 to 6.0]

4. Secondary Outcome: Heart Rate
Description: Heart rate recordings 1 minute before the first injection and at 3, 6, 9, 12, 15, 30, 45 and 60 minutes after the first injection
Time Frame: from 1 minute before to 60 minutes after the start of premedication
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Atropine + Propofol | Atropine + Atracurium + Sufentanil
Number analyzed (Participants) | 86 | 80
bpm
  Heart rate from t-1 to t+6, Difference in bpm | 3.3 (19.5) | 11.5 (19.6)
  Heart rate from t-1 to t+9, Difference in bpm | 1.6 (25.2) | 11.7 (25.3)

5. Secondary Outcome: Short Term Neurological Outcome: Worsening of Head Ultrasound
Description: Worsening of head ultrasound scans in the 7 days after intubation from the preinclusion evaluation, defined as either a normal scan before inclusion and any grade intraventricular hemorrhage (IVH) afterwards, or as a preinclusion grade 1 or 2 IVH scan deteriorating to grade 3 or 4 IVH, according to Papile's classification; This analysis was not centralized but performed in each center according to its usual protocols.
Time Frame: Within 7 days after inclusion
Measure: Count of Participants; unit: Participants
Arm/Group | Atropine + Propofol | Atropine + Atracurium + Sufentanil
Number analyzed (Participants) | 68 | 68
Participants | 14 | 12

6. Secondary Outcome: Number of Patients Surviving Without Ages and Stages Questionnaire Score Below Threshold at Age 2
Description: Survival without risk of neurodevelopmental delay. Risk of neurodevelopmental delay was defined as no Ages and Stages Questionnaires (ASQ) domain score below threshold (-2 SD) at 2 years of corrected age. The ASQ includes 30 items in 5 neurodevelopmental domains: communication abilities, gross motor skills, fine motor skills, problem solving abilities, and personal-social skills. For each domain, the score obtained by the sum of the items ranges from 0 to 60 and the overall maximum ASQ score is 300 points. For each domain, the score can be categorized using established screening thresholds: an ASQ score <-2 SD below the mean suggests a risk of neurodevelopmental delay in that domai.
Time Frame: At 2 years corrected age
Population: To handle missing data on ASQ scores, we performed multiple imputation with chained equations using the SAS "MI" procedure. The primary analysis was performed on the imputed dataset in the "as treated" study groups.
Measure: Count of Participants; unit: Participants
Groups:
- Atropine Atracurium Sufentanil "as Treated" Population: n=81
  * n=79 Received intervention as randomized
  * n=2 Allocated to atropine + propofol but did not receive propofol and received atracurium + sufentanil as open-label drug
- Atropine Propofol "as Treated" Population: n=85
  * n=83 Received intervention as randomized
  * n=1 Allocated to atropine + atracurium + sufentanil but received propofol as open-label drug
  * n=1 Allocated to atropine + propofol but did not receive intervention as randomized, received open-label atropine + propofol
Arm/Group | Atropine Atracurium Sufentanil "as Treated" Population | Atropine Propofol "as Treated" Population
Number analyzed (Participants) | 81 | 85
Participants | 38 | 45

7. Secondary Outcome: Pulse Oxymetry
Description: Pulse oxymetry recordings 1 minute before the first injection and at 3, 6, 9, 12, 15, 30, 45 and 60 minutes after the first injection
Time Frame: from 1 minute before to 60 minutes after the start of premedication
Population: Changes in SpO2 value from baseline were analyzed at predefined time points. Data was missing at some time points.
Measure: Mean (Standard Deviation); unit: % SpO2
Arm/Group | Atropine + Propofol | Atropine + Atracurium + Sufentanil
Number analyzed (Participants) | 85 | 80
% SpO2
  SpO2 from t-1 to t+6, Difference in % | -6.0 (20.1) | -12.0 (20.1)
  SpO2 from t-1 to t+9, Difference in %: number analyzed (Participants) | 84 | 80
  SpO2 from t-1 to t+9, Difference in % | -8.7 (22.3) | -15.9 (22.2)

8. Secondary Outcome: Mean Blood Pressure
Description: Blood pressure recordings 1 minute before the first injection and at 3, 6, 9, 12, 15, 30, 45 and 60 minutes after the first injection
Time Frame: from 1 minute before to 60 minutes after the start of premedication
Population: Changes from baseline in mean arterial blood pressure (MAP) were analyzed at predefined time points. Values were missing at some time points.
Measure: Mean (Standard Deviation); unit: Difference in mm Hg
Arm/Group | Atropine + Propofol | Atropine + Atracurium + Sufentanil
Number analyzed (Participants) | 80 | 77
Difference in mm Hg
  Mean arterial blood pressure from t-1 to t+15 | -6.8 (12.7) | 0.2 (12.7)
  Mean arterial blood pressure from t-1 to t+30: number analyzed (Participants) | 76 | 74
  Mean arterial blood pressure from t-1 to t+30 | -9.1 (9.3) | -3.3 (9.4)

9. Secondary Outcome: Transcutaneous PCO2 (TcPCO2) Measurement
Description: TcPCO2 recordings 1 minute before the first injection and at 3, 6, 9, 12, 15, 30, 45 and 60 minutes after the first injection
Time Frame: from 1 minute before to 60 minutes after the start of premedication
Population: Changes in TcPCO2 from baseline were analyzed at predefined time points. Values were missing at some time points.
Measure: Mean (Standard Deviation); unit: Difference in mm Hg
Arm/Group | Atropine + Propofol | Atropine + Atracurium + Sufentanil
Number analyzed (Participants) | 32 | 29
Difference in mm Hg
  TcPCO2 from t-1 to t+15 | 8.0 (14.4) | 14.1 (14.4)
  TcPCO2 from t-1 to t+30: number analyzed (Participants) | 30 | 29
  TcPCO2 from t-1 to t+30 | 5.1 (19.1) | 16.2 (19.3)

ADVERSE EVENTS:
Arm/Group | Atropine + Propofol | Atropine + Atracurium + Sufentanil
All-Cause Mortality (participants affected / at risk) | 2/83 | 3/80
Serious Adverse Events (participants affected / at risk) | 9/83 | 16/80
Other Adverse Events (participants affected / at risk) | 25/83 | 28/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atropine + Propofol (N=83) | Atropine + Atracurium + Sufentanil (N=80)
Death (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1)
Thoracic rigidity (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 11 (11)
Hypotension (treated) (Vascular disorders) | 2 (2) | 0 (0)
OTHER (General disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atropine + Propofol (N=83) | Atropine + Atracurium + Sufentanil (N=80)
Hypotension, not treated (Vascular disorders) | 9 (9) | 1 (1)
Hypertension (Vascular disorders) | 7 (7) | 7 (7)
Bradycardia (Cardiac disorders) | 1 (1) | 6 (6)
Other (General disorders) | 12 (12) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-01): https://cdn.clinicaltrials.gov/large-docs/80/NCT01490580/Prot_SAP_000.pdf